CLINICAL TRIAL: NCT00320619
Title: Aminocaproic Acid and Bleeding in Spinal Surgery
Brief Title: Epsilon-Aminocaproaic Acid to Reduce the Need for Blood Transfusions During and Following Spine Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sean Berenholtz, MD, MHS, Johns Hopkins Medical Institutions
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 360; K23HL070058-03 (NIH)
Record Dates: First submitted 2006-04-28; First posted 2006-05-03 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2009-03

CONDITIONS: Scoliosis; Kyphosis; Lordosis; Spondylitis; Spinal Stenosis
Keywords: Aminocaproic Acids; Blood Transfusion
MeSH Terms: conditions — Scoliosis; Kyphosis; Lordosis; Spondylitis; Spinal Stenosis | interventions — Aminocaproic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental): Participants will receive either EACA.
  Interventions: Drug: Epsilon-Aminocaproic Acid (EACA)
- 2 (Placebo Comparator): Participants will receive placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Epsilon-Aminocaproic Acid (EACA) — Participants will receive EACA intravenously during surgery and for 8 hours following surgery in the intensive care unit (ICU).
  Arms: 1
Drug: Placebo — Participants will receive placebo intravenously during surgery and for 8 hours following surgery in the intensive care unit (ICU).
  Arms: 2

SUMMARY:
Individuals who undergo spine surgery often have a significant loss of blood and may require multiple blood transfusions. Research has shown that epsilon-aminocaproic acid (EACA) may reduce the amount of blood lost during surgery, which would decrease the number of blood transfusions required. This study will evaluate the safety and effectiveness of EACA at reducing blood loss and the need for blood transfusions in individuals undergoing spine surgery.

DETAILED DESCRIPTION:
Spine surgery is often required to correct a number of diseases, including spondylosis, pseudoarthrosis, scoliosis, or other spinal deformities. Spine surgery is often associated with significant blood loss and individuals may require multiple blood transfusions during and following surgery. Blood transfusions are expensive and carry an increased risk of health complications, including fever, allergic reactions, or infections. Preliminary research has shown that EACA may be beneficial for individuals undergoing spine surgery. In addition, EACA appears to be safer and less expensive than other medications typically used to treat serious bleeding. The purpose of this study is to evaluate the safety and effectiveness of EACA at reducing the number of blood transfusions required during and following spine surgery in adults.

This study will enroll individuals who are undergoing spine surgery at Johns Hopkins Hospital. Prior to surgery, participants' demographic data and medical history will be collected. Participants will then be randomly assigned to receive either EACA or placebo intravenously during surgery and for 8 hours following surgery in the intensive care unit (ICU). While in the hospital, participants will have blood drawn frequently for laboratory testing. They will receive blood transfusions as needed and will be closely monitored for blood loss and any medical, surgical, or transfusion complications. Outcome measurements related to the amount of transfused blood required and postoperative complications will be collected on the 8th day following surgery. Study participation will end on the day of hospital discharge or the day of a necessary second surgery.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of spondylosis, pseudoarthrosis, kyphoscoliosis, or acquired or congenital spine deformity
* Willing to undergo elective spinal surgery by a participating surgeon; eligible procedures include the following: spine osteotomy, arthrodesis, instrumentation and/or corpectomy, surgery for lumbar spinal stenosis, or surgery for degenerative disc disease

Exclusion Criteria:

* Requires urgent or emergent surgery
* Has kidney failure that requires dialysis
* Has a known bleeding diathesis, defined as a documented history of an inherited bleeding disorder (e.g., hemophilia or von Willebrand's disease) OR prothrombin time ratio greater than 1.5 seconds OR a documented previous arterial or venous thrombosis within 1 year of study entry
* Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2000-09; Primary Completion 2006-02 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Number of allogenic blood units transfused | Measured through the 8th postoperative day

SECONDARY OUTCOMES:
Intraoperative and postoperative blood loss | Measured through the 8th postoperative day
Intraoperative and postoperative blood products received, including autologous blood, allogenic blood, fresh frozen plasma, platelets, or cryo | Measured through the 8th postoperative day
Potential complications of transfusion | Measured through the 8th postoperative day
Potential complications of EACA | Measured through the 8th postoperative day
Potential surgical complications | Measured through the 8th postoperative day
Duration of mechanical ventilation | Measured through the 8th postoperative day
In-hospital mortality | Measured through the 8th postoperative day
ICU length of stay (LOS) | Measured through the 8th postoperative day
Hospital LOS | Measured through the 8th postoperative day
Direct costs of hospital care | Measured through the 8th postoperative day

CONTACTS AND LOCATIONS:
Overall Officials: Sean Berenholtz, MD, MHS, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

REFERENCES:
- [Background] Goodnough LT, Bach RG. Anemia, transfusion, and mortality. N Engl J Med. 2001 Oct 25;345(17):1272-4. doi: 10.1056/NEJM200110253451711. No abstract available. PMID 11680450
- [Background] Troianos CA, Sypula RW, Lucas DM, D'Amico F, Mathie TB, Desai M, Pasqual RT, Pellegrini RV, Newfeld ML. The effect of prophylactic epsilon-aminocaproic acid on bleeding, transfusions, platelet function, and fibrinolysis during coronary artery bypass grafting. Anesthesiology. 1999 Aug;91(2):430-5. doi: 10.1097/00000542-199908000-00017. PMID 10443606
- [Background] Slaughter TF, Faghih F, Greenberg CS, Leslie JB, Sladen RN. The effects of epsilon-aminocaproic acid on fibrinolysis and thrombin generation during cardiac surgery. Anesth Analg. 1997 Dec;85(6):1221-6. doi: 10.1097/00000539-199712000-00008. PMID 9390584
- [Background] Florentino-Pineda I, Thompson GH, Poe-Kochert C, Huang RP, Haber LL, Blakemore LC. The effect of amicar on perioperative blood loss in idiopathic scoliosis: the results of a prospective, randomized double-blind study. Spine (Phila Pa 1976). 2004 Feb 1;29(3):233-8. doi: 10.1097/01.brs.0000109883.18015.b9. PMID 14752343
- [Derived] Berenholtz SM, Pham JC, Garrett-Mayer E, Atchison CW, Kostuik JP, Cohen DB, Nundy S, Dorman T, Ness PM, Klag MJ, Pronovost PJ, Kebaish KM. Effect of epsilon aminocaproic acid on red-cell transfusion requirements in major spinal surgery. Spine (Phila Pa 1976). 2009 Sep 1;34(19):2096-103. doi: 10.1097/BRS.0b013e3181b1fab2. PMID 19730217